CLINICAL TRIAL: NCT05818644
Title: Hepatic Artery Stenosis and Thrombosis After Liver Transplantation in Children: a Multicenter, Retrospective, Observational Study
Brief Title: Hepatic Artery Stenosis and Thrombosis After Liver Transplantation in Children
Acronym: HEPATIC
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: J. P. Garrahan Hospital (Unknown); Hospital Italiano de Buenos Aires (Other); Royal Children's Hospital (Other); Medical University of Innsbruck (Unknown); Hospital Sírio-Libanês (Unknown); Hospital Santo Antonio (Unknown); Faculty of Medicine & Dentistry, University of Alberta (Unknown); Zhejiang University (Other); Thomayer University Hospital (Other); Hôpital Bicêtre (Unknown); University Children's Hospital (Other); Hannover Medical School (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Dr Rela Institute and Medical Centre (Unknown); Amrita Institute of Medical Sciences & Research Centre (Unknown); Max Super Speciality Hospital (Other); Aster CMI Hospital (Unknown); ASST Papa Giovanni XXIII Hospital (Unknown); Bambino Gesù Children's Hospital (Unknown); National Centre for Child Health and Development (Unknown); Auckland City Hospital (Other Government); Children's Memorial Health Institute (Unknown); King Faisal Specialist Hospital & Research Center (Other); National University Hospital, Singapore (Other); Wits Donald Gordon Medical Centre (Unknown); La Paz University Hospital (Unknown); Vall d'Hebron Barcelona Hospital Campus (Unknown); Karolinska Institutet (Other); University Hospital, Geneva (Other); Birmingham Women's and Children's Hospital (Unknown); Primary Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Pittsburgh (Unknown); Recanati-Miller Transplantation Institute, Mount Sinai Hospital (Unknown); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 17033
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Hepatic Artery Thrombosis; Hepatic Artery Stenosis; Pediatric ALL; Liver Transplant; Complications
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Conservative treatment
- Surgical revascularization
- Endovascular revascularization
- Re-transplantation

SUMMARY:
The goal of this observational study is to investigate the incidence, current management practices, and outcomes in pediatric patients with HAC after liver transplantation.

Research question:

* What are the overall incidence of HAC and the effectiveness of all treatment strategies for HAC after pediatric LT?
* What are the current management practices in the experience of centers, anticoagulant therapy, screening protocol, and assessment criteria for HAC after pediatric LT?

The burden of participation is considered to be minimal, and limited to the questionnaires.

ELIGIBILITY:
Inclusion criteria:

* Liver transplantation between January 1st 2002 and January 1st 2022, diagnoses of HAC after LT
* The age of the patient is below 18 years at the time of diagnosis and intervention
* The date of diagnosis of HAC or intervention was before January 1st 2023. HAC occurring after first or subsequent LTs are included.

Exclusion criteria:

N/A

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any pediatric patient diagnosed with HAC and treated for HAC (at age <18 years) after pediatric liver transplantation between 1-1-2002 and 1-1-2023
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Graft survival | 1-1-2001 and 1-1-2023
  Graft survival is defined as a functioning graft from transplantation to the end of follow-up data, re-transplantation, or death, whichever occurs first.
Patient survival | 1-1-2001 and 1-1-2023
  Patient survival is defined from the date of the primary LT until date of death. Causes of re-transplantation or death will be recorded.

SECONDARY OUTCOMES:
Technical success | 1-1-2001 and 1-1-2023
  Technical success is defined as the success of the intervention in re-establishing the arterial blood flow to the liver and will be assessed by each individual center.
Primary and secondary patency | 1-1-2001 and 1-1-2023
  Primary patency is defined as the time between the index treatment and re-intervention intended to restore patency in patients with a restenosis or re-occlusion. Secondary patency is the time between the index treatment and failure to re-establish flow by means of re-intervention. In case of re-transplantation or death due to other reasons, the patients will be censored if the treated vessel is patent. Kaplan-Meier curves will be plotted to visualize primary and secondary patency rates at various times after treatment for HAC, including 1, 3, 5, 10, 15 and 20 years.
Intra- and post-procedural complications | 1-1-2001 and 1-1-2023
  Procedural complications will be categorized into two main groups: transplant complications and procedural complications related to endovascular or surgical revascularization for HAC. Within these groups, intra-procedural complications predominantly consist of vascular issues, such as thrombosis, stenosis, compression, dissection, and rupture. In contrast, post-procedural complications encompass a broader range of issues, such as infection, rejection, bleeding, and vascular and biliary complications, including anastomotic stricture, non-anastomotic strictures, bile leak, biloma, or cholangitis. Re-interventions addressing both intra- and post-procedural complications will also be recorded.
Anticoagulant therapy after transplantation and after interventions | 1-1-2001 and 1-1-2023
  Anticoagulant therapy after transplantation and after interventions for HAC will be assessed according to the management practices of each participating site (center specific) and individual patient data (patient specific). Details about each anticoagulation regimen, including the specific anticoagulant, duration of anticoagulation, and upper and lower limits of target values, such as international normalized ratio, anti-factor Xa, and activated partial thromboplastin time, will be recorded. Patient-specific management will be documented for patients with HAC.
Center specific screening protocol | 1-1-2001 and 1-1-2023
  Local screening protocols to assess HAC after LT, such as the routine post-operative Doppler ultrasound policy, will be documented. Whether HAC screening is consistent for patients with and without risk factors will also be examined. The frequency of preferred radiological screening investigations within 2 weeks after LT will be determined, considering various risk factors.
Center specific diagnostic criteria | 1-1-2001 and 1-1-2023
  The diagnostic criteria section will cover the types of HAC, non-invasive radiological criteria, and interventional radiological criteria during invasive angiography. The center's definition of technical success after interventional radiological treatment will also be recorded.
Center specific radiological follow up | 1-1-2001 and 1-1-2023
  The radiological follow-up section will assess whether follow-up protocols are the same for all interventions or specific to each intervention type. The imaging methods and frequencies of radiological follow-up for different treatment modalities will be determined. Additionally, the experience years and level of seniority of the interventional radiologist will be recorded.
Incidence | 1-1-2001 and 1-1-2023
  The incidence of HAC will be determined by dividing the total number of patients diagnosed with HAC between 1st of January 2002 and 1st of January 2023, who had undergone LT between 1st of January 2002 and 1st of January 2022, by the total number of patients who underwent LT at pediatric age between 1st of January 2002 and 1st of January 2022. The study will present the overall incidence of HAC during the 20-year period of 2002 to 2022, as well as the incidence during specific 5-year intervals, namely 2002 to 2007, 2007 to 2012, 2012 to 2017, and 2017 to 2022, for each complication.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li W, van der Doef HPJ, Wildhaber BE, Marra P, Bravi M, Pinelli D, Minetto J, Dip M, Sierre S, de Santibanes M, Ardiles V, Uno JW, Hardikar W, Bates S, Goh L, Aldrian D, Seisenbacher J, Vogel GF, Neto JS, Antunes da Fonseca E, Magalhaes Costa C, Ferreira CT, Nader LS, Farina MA, Dajani KZ, Parente A, Bigam DL, Liang TB, Bai X, Zhang W, Gonsorcikova L, Fronek J, Bohus S, Franchi-Abella S, Gonzales E, Guerin F, Junge N, Baumann U, Richter N, Hartleif S, Sturm E, Rajakannu M, Palaniappan K, Rela M, Pawaria A, Rajakrishnan H, Surendran S, Kumar M, Agarwal S, Gupta S, Asthana S, Bandewar V, Raichurkar K, Spada M, Monti L, Alterio T, Yanagi Y, Uchida H, Komine R, Evans H, Carr-Boyd P, Duncan D, Stefanowicz M, Latka-Grot J, Kolesnik A, Broering DC, Raptis DA, Ann H Marquez K, Mali V, Aw M, Beretta M, Van der Schyff F, Quintero-Bernabeu J, Mercadal-Hally M, Larrarte K M, Andres AM, Hernandez-Oliveros F, Frauca E, Casswall T, Jorns C, Delle M, Gupte G, Sharif K, McGuirk S, Superina R, Caicedo JC, Jaramillo C, Bitterfeld L, Kastenberg Z, Shah AA, Domenick B, Acord MR, Mazariegos GV, Soltys K, DiNorcia J, Antala S, Florman SS, Buchholz BM, Herden U, Fischer L, Dierckx RAJO, Hartog H, Bokkers RPH. Incidence, management and outcomes in hepatic artery complications after paediatric liver transplantation: protocol of the retrospective, international, multicentre HEPATIC Registry. BMJ Open. 2024 Jun 12;14(6):e081933. doi: 10.1136/bmjopen-2023-081933. PMID 38866577